CLINICAL TRIAL: NCT02789371
Title: Comparing of Modified Wet Suction Technique and Dry Suction Technique for Endoscopic Ultrasound -Guided Fine Needle Aspiration (EUS-FNA) of Solid Occupying Lesions: a Prospective Multi-center,Randomized,and Controlled Trial
Brief Title: Comparing of Modified Wet Suction Technique and Dry Suction Technique for EUS-FNA of Solid Occupying Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bin Cheng (Other)
Responsible Party: Sponsor-Investigator, Bin Cheng, professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: S135
Record Dates: First submitted 2016-05-21; First posted 2016-06-03 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Pancreas Neoplasms; Lymphatic Metastasis; Neoplasm Metastases; Unknown Primary Neoplasm Metastasis; Infection; Inflammation; Sarcoid; Lymphadenopathy
Keywords: EUS-FNA; modified wet suction technique; dry suction technique
MeSH Terms: conditions — Pancreatic Neoplasms; Lymphatic Metastasis; Neoplasm Metastasis; Neoplasms, Unknown Primary; Infections; Inflammation; Sarcoidosis; Lymphadenopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Other): the first pass is made with 5ml suction technique
  Interventions: Procedure: the first pass is made with 5ml suction technique
- Arm B (Other): the first pass is made with modified wet suction technique
  Interventions: Procedure: the first pass is made with modified wet suction technique

INTERVENTIONS:
Procedure: the first pass is made with 5ml suction technique — the first pass is made with 5ml suction technique, then modified wet suction technique / 5ml suction technique/ modified wet suction technique is operated successively.
  Arms: Arm A
Procedure: the first pass is made with modified wet suction technique — the first pass is made with modified wet suction technique, then 5ml suction technique/ modified wet suction technique/ 5ml suction technique is operated successively.
  Arms: Arm B

SUMMARY:
The purpose of this study is to compare the diagnosis accuracy of modified wet suction technique and 5ml dry suction technique on solid occupying lesions.

DETAILED DESCRIPTION:
Patients will be divided into two groups, arm A and arm B according to two different methods adopted in their first needle, which refers to the modified wet suction technique or 5ml dry suction technique.Take the solid occupying lesion diagnosis accuracy as the research major indicator to compare the the modified wet suction technique or 5ml dry suction technique as optimal efficiency test. Take classⅠerror, a=0.05, class II error, β=0.2, power=0.8, suppose that the diagnostic accuracy of dry suction technique to the solid occupying lesions is 75%, the diagnostic accuracy of modified wet suction technique to the solid occupying lesions is 85%, the minimum sample size are 248 patients with 5ml dry suction technique and 248 patients with modified wet suction technique, the 2x2 cross-over design is adopted, namely, each arm has 124 patients respectively. Considering factors including defluxion, 20% cases will be added to two arms, therefore, each arm has 148 patients respectively, the total number of patients is 296.

The statistics experts generated randomized serial numbers（001-296）according to same-size allocation ratio between arm A and arm B with Statistical Analysis System 9.2(SAS 9.2), a statistical software in the randomized block method. The serial numbers are the randomized grouping numbers for the trial patients, block capacity is 8, totally 37 randomized block. One copy send to trial centers for patient allocating, and the another copy be saved by the trial applicant unit. Every trail centers will be responsible for the screening of qualified patients, rank them in visit time to get the randomized grouping number so as to determine them goes to arm A or arm B .The research people and patients in all trial centers should not know the randomized grouping number and relevant arms. The arm name will be sealed under scratch card. Every trial patients will get a unique randomized number, and it will not change through out the whole trial.

Use the inclusion and exclusion criteria to observe the patients and do relative inspections, and confirm if the patients qualified or not to the trial. Record the result of last time test before the treatment. Although it is better to get the informed consent before doing all kinds of observation and tests, if for some reason, the medical imaging examination has completed,as long as the imaging examination was done within 3 weeks before the needle biopsy, it can still be collect as baseline data (imaging examination can be done at other hospitals, but the trial center should issue a new evaluation report 1 week before the patient join the trial group); other lab test items done at 2 weeks before the needle biopsy can still be collect as baseline data for pre-research use, but these tests should be done at the trail center hospital so as to guarantee the data trace ability.

The investigator will puncture the lesion for four needle passes for all of them:For Arm A,5ml dry suction technique is adopted in their first needle, then modified wet suction technique/5ml dry suction technique/modified wet suction technique is operated successively;For Arm B, modified wet suction technique is adopted in their first needle, then 5ml dry suction technique/ modified wet suction technique /5ml dry suction technique is operated successively.Well,the 5ml dry suction technique is conducted as follow:after the needle puncturing into the lesion under ultrasound scanning, remove the stylet and connect the needle to syringe with 5ml negative pressure aspiration, then the needle will be moved to-and-fro within the lesion 20 times. Suction will be released before the needle is withdrawn from the lesion.And the modified wet suction technique is conducted as follow:the needle whose stylet is pulled out will be flushed with 2ml saline solution before puncturing when the lesion has been found, then puncture into the lesions and replace syringe with 5ml negative pressure aspiration, then the needle will be moved to-and-fro within the lesion 20 times. Suction will be released before the needle is withdrawn from the lesion.If no core tissues obtained or the operator determine insufficient specimen according to Macroscopic rapid on-site(MOSE) after the operations above, then remedy procedures will be done, and the punctuation process should be continued with the appropriate punctuation methods until the satisfactory specimens are obtained.Experts in cytology and pathology evaluate the specimen quality and make a diagnosis under the condition that they do not know punctuation methods. The evaluation and diagnosis of each specimen are made by two experts independently. If the two experts hold different opinions, they will make a conclusion after full discussion. If there are two or more cytological smears with same punctuation method, the highest-rate smear should be taken as the standard smear.Follow up (outpatient follow up or telephone follow up) the patients at 1 week, 12 weeks and 36 weeks after the needle biopsy and collect the patients clinical data and confirm their final diagnosis.

Case Report Form(CRF) will be filled by the researchers, every involved patient must have the CRF filled. This will be audited by clinical monitor and handed over to data administrator to input and manage data, the first copy will be kept by the applicant, the second copy will go to the trial center, and the third copy will be kept by the trail researchers.The data input and management will be taken care by specially assigned person. In order to guarantee the data accuracy, data input will be done twice by two independent data administrators, by computerized and manual verifying, hand over the data to statistical experts to do blind check and statistic analyzing.For the questions and doubts within the case report form, the data administrator make DRQ and via the clinical monitor asking the researchers. The researchers will answer and feed back as soon as possible. According to the researchers answer, data administrator will do the data modifying, confirming or inputting, and when necessary send out DRQ again.After blind audition and confirming that the established data base is correct, major researchers, applicant and the statistic analyzing people lock the data. The locked data will not be changed, and the data base will be handed over to statistical analyzer to do the statistic analyze according to the statistic analyzing plan. Problems found after data locking can be modified during the statistic analyzing procedure.This will be done by specialized statistic analyzing people according to the predetermined statistic analyzing plan. The statistic analyze will be carried out according to intention principle confirmed full analysis set and per-protocol set principle. After completing the statistic analyzing, the statistic analyzer issue the statistic analysis report and send this to major researchers to write the study report.

Statistic analyzing plan:（1）General principle①All statistical tests were two-sided. P<0.05 is regarded that the difference is statistical significance.② Description of quantitative index will calculate the mean and the criteria deviation, description of classification index will describe the number and percentage of each type.（2） Statistical Analysis Method：① For measurement data, compare these data with baseline value during the screening period, adopt the deviation t-test, the variance analysis of cross-over experiment or the rank-sum test of cross-over experiment to make a comparison between these data and baseline value.② For enumeration data, adopt the paired x2-test(including CMH-x2 test) or Fisher's exact test to compare these data of each group.（3）Defluxion Analysis：The total defluxion rate of each group and the defluxion rate caused by adverse events are compared by x2-test or Fisher's exact test.（4）Analysis of baseline value balance：The indexes of some baseline values such as demographic data, vital signs, history of diseases and basic treatment are compared by group t-test and x2 test to measure the balance of each group. Baseline evaluation is made to full analysis set( FAS) and per-protocol set(PPS).（5）Validity Analysis：The primary index of validity analysis is the diagnostic accuracy of the 5ml dry pressure and modified wet pressure to the solid space-occupying lesions. The secondary indexes of validity analysis include the punctuation specimen quality of 5ml dry pressure and modified wet pressure, the diagnostic rate of the first needle of 5ml dry pressure / modified wet pressure and the incidence of complications for modified wet pressure and 5ml dry pressure. The rates of each two arms and Youden indexes are compared by the approximate normal z-test or the central-effect-considered Cochran Mantel Haenszel-x2(CMH-x2 )text.(6)Safety Analysis:The incidences of adverse events/ adverse reactions (including complications from punctuation) of each arm are compared by x2-test or Fisher's exact test and describe the adverse events occurred in this experiment by the list and the normal/abnormal changes of laboratory text results before and after test and the relationship between abnormal changes of laboratory text results and this diagnostic research.(7) All statistical analyses are completed by the professional statistical analysis software, SAS version 9.2.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old,<80 years old;
2. Gender: Male or Female;
3. The patients who have solid occupying pancreatic lesions and non-pancreatic lesions (the diameter>1cm) within the range of imaging examination(MRI、CT、B-type ultrasonography) and ultrasonic endoscope examination and should conduct the biopsy to identify lesion nature;
4. The patients who receive examinations in the research center;
5. The patients who sign the informed consent.

Exclusion Criteria:

1. Hemoglobin≤8.0 g/dl;
2. Pregnant women;
3. The patients who have coagulation disorders（PLT<50,000/mm3,INR>1.5,roughly calculation, INR>1.5, is equivalent to PT>18 seconds);
4. The patients who took anticoagulants such as aspirin, warfarin in the latest week;
5. The patients who suffered from acute pancreatitis in the past two weeks;
6. The patients who have cardiopulmonary dysfunction, therefore cannot tolerate ultrasonic endoscope examination;
7. The patients who cannot sign the informed consent(such as patients who have mental disease or drug addiction and so on).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-02 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
the overall diagnostic accuracy of modified wet suction technique and 5ml dry suction technique to the solid occupying lesions | 18 months
  The investigators' primary outcome measure is to compare the overall diagnostic accuracy of modified wet suction technique and dry suction technique to the solid occupying lesions.

SECONDARY OUTCOMES:
the diagnostic accuracy of modified wet suction technique and 5ml dry suction technique to the benign and malignant solid occupying pancreatic lesions and non-pancreatic lesions respectively. | 18 months
  The investigators'secondary outcome measure is to compare the diagnostic accuracy of modified wet suction technique and 5ml dry suction technique to the benign and malignant solid occupying pancreatic lesions and non-pancreatic lesions respectively.
Blood contamination and cellularity in specimens obtained by modified wet suction technique and 5ml dry suction technique | 18 months
  The investigators'secondary outcome measure is to compare the cellularity and blood cell contamination of the solid occupying lesions with modified wet suction technique and 5ml dry suction technique.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cheng, Doctor, Principal Investigator — Tongji Hospital; Yun Wang, Doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Furukawa H, Okada S, Kakizoe T. Early diagnosis of pancreatic cancer. Hepatogastroenterology. 1999 Jan-Feb;46(25):4-7. PMID 10228757
- [Result] Furukawa H, Okada S, Saisho H, Ariyama J, Karasawa E, Nakaizumi A, Nakazawa S, Murakami K, Kakizoe T. Clinicopathologic features of small pancreatic adenocarcinoma. A collective study. Cancer. 1996 Sep 1;78(5):986-90. doi: 10.1002/(SICI)1097-0142(19960901)78:53.0.CO;2-A. PMID 8780535
- [Result] DeWitt J, Jowell P, Leblanc J, McHenry L, McGreevy K, Cramer H, Volmar K, Sherman S, Gress F. EUS-guided FNA of pancreatic metastases: a multicenter experience. Gastrointest Endosc. 2005 May;61(6):689-96. doi: 10.1016/s0016-5107(05)00287-7. PMID 15855973
- [Result] Puli SR, Batapati Krishna Reddy J, Bechtold ML, Ibdah JA, Antillon D, Singh S, Olyaee M, Antillon MR. Endoscopic ultrasound: it's accuracy in evaluating mediastinal lymphadenopathy? A meta-analysis and systematic review. World J Gastroenterol. 2008 May 21;14(19):3028-37. doi: 10.3748/wjg.14.3028. PMID 18494054
- [Result] Gress FG, Hawes RH, Savides TJ, Ikenberry SO, Lehman GA. Endoscopic ultrasound-guided fine-needle aspiration biopsy using linear array and radial scanning endosonography. Gastrointest Endosc. 1997 Mar;45(3):243-50. doi: 10.1016/s0016-5107(97)70266-9. PMID 9087830
- [Result] Savides TJ, Donohue M, Hunt G, Al-Haddad M, Aslanian H, Ben-Menachem T, Chen VK, Coyle W, Deutsch J, DeWitt J, Dhawan M, Eckardt A, Eloubeidi M, Esker A, Gordon SR, Gress F, Ikenberry S, Joyce AM, Klapman J, Lo S, Maluf-Filho F, Nickl N, Singh V, Wills J, Behling C. EUS-guided FNA diagnostic yield of malignancy in solid pancreatic masses: a benchmark for quality performance measurement. Gastrointest Endosc. 2007 Aug;66(2):277-82. doi: 10.1016/j.gie.2007.01.017. PMID 17643700
- [Result] Sadeghi A, Mohamadnejad M, Islami F, Keshtkar A, Biglari M, Malekzadeh R, Eloubeidi MA. Diagnostic yield of EUS-guided FNA for malignant biliary stricture: a systematic review and meta-analysis. Gastrointest Endosc. 2016 Feb;83(2):290-8.e1. doi: 10.1016/j.gie.2015.09.024. Epub 2015 Sep 28. PMID 26422979
- [Result] Lee JK, Choi JH, Lee KH, Kim KM, Shin JU, Lee JK, Lee KT, Jang KT. A prospective, comparative trial to optimize sampling techniques in EUS-guided FNA of solid pancreatic masses. Gastrointest Endosc. 2013 May;77(5):745-51. doi: 10.1016/j.gie.2012.12.009. Epub 2013 Feb 21. PMID 23433878
- [Result] Ogura T, Yamao K, Sawaki A, Mizuno N, Hara K, Hijioka S, Niwa Y, Tajika M, Kondo S, Shimizu Y, Bhatia V, Higuchi K, Hosoda W, Yatabe Y. Clinical impact of K-ras mutation analysis in EUS-guided FNA specimens from pancreatic masses. Gastrointest Endosc. 2012 Apr;75(4):769-74. doi: 10.1016/j.gie.2011.11.012. Epub 2012 Jan 28. PMID 22284089
- [Result] Iglesias-Garcia J, Poley JW, Larghi A, Giovannini M, Petrone MC, Abdulkader I, Monges G, Costamagna G, Arcidiacono P, Biermann K, Rindi G, Bories E, Dogloni C, Bruno M, Dominguez-Munoz JE. Feasibility and yield of a new EUS histology needle: results from a multicenter, pooled, cohort study. Gastrointest Endosc. 2011 Jun;73(6):1189-96. doi: 10.1016/j.gie.2011.01.053. Epub 2011 Mar 21. PMID 21420083
- [Result] Puri R, Vilmann P, Saftoiu A, Skov BG, Linnemann D, Hassan H, Garcia ES, Gorunescu F. Randomized controlled trial of endoscopic ultrasound-guided fine-needle sampling with or without suction for better cytological diagnosis. Scand J Gastroenterol. 2009;44(4):499-504. doi: 10.1080/00365520802647392. PMID 19117242
- [Result] Attam R, Arain MA, Bloechl SJ, Trikudanathan G, Munigala S, Bakman Y, Singh M, Wallace T, Henderson JB, Catalano MF, Guda NM. "Wet suction technique (WEST)": a novel way to enhance the quality of EUS-FNA aspirate. Results of a prospective, single-blind, randomized, controlled trial using a 22-gauge needle for EUS-FNA of solid lesions. Gastrointest Endosc. 2015;81(6):1401-7. doi: 10.1016/j.gie.2014.11.023. Epub 2015 Feb 27. PMID 25733127
- [Result] Villa NA, Berzosa M, Wallace MB, Raijman I. Endoscopic ultrasound-guided fine needle aspiration: The wet suction technique. Endosc Ultrasound. 2016 Jan-Feb;5(1):17-20. doi: 10.4103/2303-9027.175877. PMID 26879162
- [Result] Iwashita T, Nakai Y, Samarasena JB, Park DH, Zhang Z, Gu M, Lee JG, Chang KJ. High single-pass diagnostic yield of a new 25-gauge core biopsy needle for EUS-guided FNA biopsy in solid pancreatic lesions. Gastrointest Endosc. 2013 Jun;77(6):909-15. doi: 10.1016/j.gie.2013.01.001. Epub 2013 Feb 20. PMID 23433596
- [Result] Fabbri C, Luigiano C, Maimone A, Tarantino I, Baccarini P, Fornelli A, Liotta R, Polifemo A, Barresi L, Traina M, Virgilio C, Cennamo V. Endoscopic ultrasound-guided fine-needle biopsy of small solid pancreatic lesions using a 22-gauge needle with side fenestration. Surg Endosc. 2015 Jun;29(6):1586-90. doi: 10.1007/s00464-014-3846-6. Epub 2014 Oct 11. PMID 25303907
- [Result] Alatawi A, Beuvon F, Grabar S, Leblanc S, Chaussade S, Terris B, Barret M, Prat F. Comparison of 22G reverse-beveled versus standard needle for endoscopic ultrasound-guided sampling of solid pancreatic lesions. United European Gastroenterol J. 2015 Aug;3(4):343-52. doi: 10.1177/2050640615577533. PMID 26279842
- [Result] Layfield LJ, Schmidt RL, Hirschowitz SL, Olson MT, Ali SZ, Dodd LL. Significance of the diagnostic categories "atypical" and "suspicious for malignancy" in the cytologic diagnosis of solid pancreatic masses. Diagn Cytopathol. 2014 Apr;42(4):292-6. doi: 10.1002/dc.23078. Epub 2014 Feb 28. PMID 24578254
- [Result] Nguyen TQ, Kalade A, Prasad S, Desmond P, Wright G, Hart D, Conron M, Chen RY. Endoscopic ultrasound guided fine needle aspiration (EUS-FNA) of mediastinal lesions. ANZ J Surg. 2011 Jan;81(1-2):75-8. doi: 10.1111/j.1445-2197.2010.05266.x. PMID 21299803
- [Derived] Wang Y, Wang RH, Ding Z, Tan SY, Chen Q, Duan YQ, Zhu LR, Cao JW, Wang J, Shi G, Wu XL, Wang JL, Zhao YC, Tang SJ, Cheng B. Wet- versus dry-suction techniques for endoscopic ultrasound-guided fine-needle aspiration of solid lesions: a multicenter randomized controlled trial. Endoscopy. 2020 Nov;52(11):995-1003. doi: 10.1055/a-1167-2214. Epub 2020 May 15. PMID 32413915
- [Derived] Wang Y, Chen Q, Wang J, Wu X, Duan Y, Yin P, Guo Q, Hou W, Cheng B. Comparison of modified wet suction technique and dry suction technique in endoscopic ultrasound-guided fine-needle aspiration (EUS-FNA) for solid lesions: study protocol for a randomized controlled trial. Trials. 2018 Jan 17;19(1):45. doi: 10.1186/s13063-017-2380-y. PMID 29343303